CLINICAL TRIAL: NCT02427659
Title: High Technology Pain Control During Burn Wound Care
Brief Title: VR High Tech Pain Control Burn Wound Care
Acronym: VRH2O
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, David R. Patterson, Professor, National Institute of General Medical Sciences (NIGMS)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 41673
Record Dates: First submitted 2015-03-31; First posted 2015-04-28 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Pain; Burn
Keywords: VRD; Virtual Reality as Distraction during Procedure; Burn Wound Care
MeSH Terms: conditions — Pain; Burns

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Virtual Reality Distraction (Other): The subjects will receive a 20-minute Virtual Reality Distraction (VRD) during their wound care procedure. The nurse will be doing their wound care.
  Interventions: Behavioral: Virtual Reality Distraction
- Audio (sounds of nature) (Other): The subjects will listen to an audio recording called "Sounds of Nature" during their wound care. The nurse will be doing the wound care.
  Interventions: Behavioral: Audio (sound of nature)
- control standard nurse wound care (Other): The subjects will receive their standard care during wound care. The nurse will be doing the wound care.
  Interventions: Behavioral: Control standard nurse wound care

INTERVENTIONS:
Behavioral: Virtual Reality Distraction — The subjects will receive a 20-minute Virtual Reality Distraction (VRD) during their wound care procedure. The nurse will be doing their wound care.
  Other Names: VRD
  Arms: Virtual Reality Distraction
Behavioral: Audio (sound of nature) — The subjects will listen to an audio recording called "Sounds of Nature" during their wound care.
  Arms: Audio (sounds of nature)
Behavioral: Control standard nurse wound care — The subjects will receive their standard care during wound care. The nurse will be doing the wound care.
  Arms: control standard nurse wound care

SUMMARY:
Using virtual reality as a form of distraction for pain during wound care. Virtual reality involves looking into a set of goggles and then moving through a computer-simulated world.

DETAILED DESCRIPTION:
This study has three different groups. Patients will be randomly assigned to one of three groups (two treatments and one control). Treatment for Group 1 is Virtual Reality Distraction during wound care. Group 2 will listen to an audio recording called "Sounds of Nature". Group 3 will be the control group.

Subjects in all three groups will receive the following questionnaires:

Graphic Rating Scale McGill Short-Form pain questionnaire Sullivan Catastrophization scale (only on Day 1/Baseline) The Nurse GRS

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Compliant and able to complete questionnaires
* No history of psychiatric disorder
* Not demonstrating delirium, psychosis or any form of Organic Brain Disorder
* Able to communicate verbally
* English-speaking

Exclusion Criteria:

* Age less than 18 years
* Not capable of indicating pain intensity
* Not capable of filling out study measures
* Evidence of traumatic brain injury
* History of psychiatric disorder
* Demonstrating delirium, psychosis or any form of Organic Brain Disorder and associated memory problems
* Unable to communicate orally
* Receiving prophylaxis for alcohol or drug withdrawal
* Developmental disability
* Any face/head/neck injuries that interfere with the use of Virtual Reality equipment
* Non-English Speaking
* Extreme susceptibility to motion sickness
* Seizure history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-11; Primary Completion 2016-11 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
"Pain" as measured by McGill Short Form Pain Questionnaire | up to an hour
  Pain is being measured
"Pain" as measured by Nurse Graphic Rating Scale | up to 3 hours
  Pain is being measured.
"Pain and anxiety" as measured by Graphic Rating Scale | up to an hour
  Pain and anxiety is being measured

CONTACTS AND LOCATIONS:
Overall Officials: David R. Patterson, Ph.D., Principal Investigator — University fo Washington
Locations (1):
- University of Washington; Harborview Medical Center, Seattle, Washington, United States